CLINICAL TRIAL: NCT02595307
Title: Role of a Written Summary on Risk Recall During Consent Process for Cleft Palate Repair
Brief Title: Improving Informed Consent for Cleft Palate Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IWK Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1015947
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Cleft Palate; Jaw Abnormalities; Maxillofacial Abnormalities; Mouth Abnormalities; Congenital Abnormalities; Jaw Diseases; Musculoskeletal Diseases; Craniofacial Abnormalities; Musculoskeletal Abnormalities; Stomatognathic Diseases; Stomatognathic System Abnormalities
Keywords: Risk Recall; Pamphlet; Brochure; Patient satisfaction; Informed Consent
MeSH Terms: conditions — Cleft Palate; Jaw Abnormalities; Maxillofacial Abnormalities; Mouth Abnormalities; Congenital Abnormalities; Jaw Diseases; Musculoskeletal Diseases; Craniofacial Abnormalities; Musculoskeletal Abnormalities; Stomatognathic Diseases; Stomatognathic System Abnormalities; Patient Satisfaction

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Pamphlet (Experimental): Participant group that will receive a written pamphlet outlining the risks of surgery as discussed in consultation.
  Interventions: Behavioral: Pamphlet
- No Pamphlet (No Intervention): Patient group that will not receive a written pamphlet outlining the risks of surgery as discussed in consultation.

INTERVENTIONS:
Behavioral: Pamphlet — Written pamphlet outlining the risks of surgery as discussed in consultation.
  Arms: Pamphlet

SUMMARY:
To determine if providing a written document in addition to the standard oral discussion of surgical risks improves risk recall for the parents/guardians of a child seen in consultation for cleft palate surgery, and if this has any effect on overall satisfaction after the procedure

DETAILED DESCRIPTION:
The current standard of care as it relates to informed consent in the pediatric population involves providing the parents or guardians of the child undergoing surgery with an oral discussion prior to the surgical procedure. However, providing parents with an oral discussion alone may be insufficient in the informed consent process as it has been shown that oral information tends to be retained poorly and crucial pieces of information tend to be forgotten. Conversely, it has been shown that properly informed patients are more satisfied, have a higher commitment to their treatment, and demonstrate less tendency toward filing legal claims. Furthermore, written material may help reduce anxiety in patients facing stressful events, such as surgery, and have been linked with overall improvement in satisfaction with their treatment

The investigators hypothesize that providing a written document in conjunction with the standard oral discussion improves the participants' risk recall in the informed consent process for their child's cleft palate repair surgery and increases their subjective satisfaction with the operation.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardians of a child referred to the IWK Cleft Palate Clinic for primary cleft palate repair surgery

Exclusion Criteria:

* Inability to fluently communicate in English
* Inability to read at a grade 8 level
* Inability to provide informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of risks recalled | 3 weeks
  The number of risks that are recalled by the patient at a 3 week follow up phone call.

SECONDARY OUTCOMES:
Participant Satisfaction as measured with the visual-analogue scale | 3 months
  Participants' perceived satisfaction with the procedure as measured with the visual-analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bezuhly, MD FRCSC, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Center, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Aggregate results only will be shared.

REFERENCES:
- [Background] Aremu SK, Alabi BS, Segun-Busari S. The role of informed consent in risks recall in otorhinolaryngology surgeries: verbal (nonintervention) vs written (intervention) summaries of risks. Am J Otolaryngol. 2011 Nov-Dec;32(6):485-9. doi: 10.1016/j.amjoto.2010.09.012. Epub 2010 Nov 19. PMID 21093107
- [Background] Nadeau DP, Rich JN, Brietzke SE. Informed consent in pediatric surgery: Do parents understand the risks? Arch Otolaryngol Head Neck Surg. 2010 Mar;136(3):265-9. doi: 10.1001/archoto.2010.5. PMID 20231645
- [Background] Lavelle-Jones C, Byrne DJ, Rice P, Cuschieri A. Factors affecting quality of informed consent. BMJ. 1993 Apr 3;306(6882):885-90. doi: 10.1136/bmj.306.6882.885. PMID 8490411
- [Background] Leclercq WK, Keulers BJ, Houterman S, Veerman M, Legemaate J, Scheltinga MR. A survey of the current practice of the informed consent process in general surgery in the Netherlands. Patient Saf Surg. 2013 Jan 21;7(1):4. doi: 10.1186/1754-9493-7-4. PMID 23336609
- [Background] Leclercq WK, Keulers BJ, Scheltinga MR, Spauwen PH, van der Wilt GJ. A review of surgical informed consent: past, present, and future. A quest to help patients make better decisions. World J Surg. 2010 Jul;34(7):1406-15. doi: 10.1007/s00268-010-0542-0. PMID 20372902
- [Background] Chan Y, Irish JC, Wood SJ, Rotstein LE, Brown DH, Gullane PJ, Lockwood GA. Patient education and informed consent in head and neck surgery. Arch Otolaryngol Head Neck Surg. 2002 Nov;128(11):1269-74. doi: 10.1001/archotol.128.11.1269. PMID 12431168
- [Background] Siau D, List RJ, Hussin N, Woolford TJ. Do printed information leaflets improve recall of the procedure and risks in adult tonsillectomy? How we do it. Clin Otolaryngol. 2010 Dec;35(6):503-6. doi: 10.1111/j.1749-4486.2010.02227.x. No abstract available. PMID 21199416